CLINICAL TRIAL: NCT03383510
Title: An Intervention Study of Sustainable Food Habits That Promotes Health and Environmental Aspects
Brief Title: Climate Friendly and Ecological Food on Microbiota
Acronym: CLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mälardalen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017/306
Record Dates: First submitted 2017-09-29; First posted 2017-12-26 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Sustainability; Microbiota; Pesticides; Organic Food
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Climate friendly group (Experimental): The climate friendly group will receive instructions to eat according to a climate friendly diet, i.e., to replace the majority of their intake of animal based products with plant based food.
  Interventions: Other: Climate friendly diet
- Organic group (Experimental): The organic group will receive instructions to eat an organic diet, i.e., to replace at least 50% of their normally consumed food with organic equivalents.
  Interventions: Other: Organic diet
- Climate friendly and organic group (Experimental): The climate friendly and organic group will receive instructions to consume a climate friendly and organic diet, i.e, to replace the majority of their intake of animal based products with plant based food AND to consume at least 50% organic food products.
  Interventions: Other: Climate friendly and organic diet
- Control group (Placebo Comparator): The control group will receive instructions to eat according to the Nordic Nutrition Recommendations.
  Interventions: Other: Control group (Control diet)

INTERVENTIONS:
Other: Climate friendly diet — Participants in the 'Climate friendly' group will be assigned a diet generating low emissions of greenhouse gases. The target is to reduce the participants' diet-related carbon dioxide equivalents (CO2e) to 2.5 kg per person and day, which is approximately a reduction by 50% compared the average CO2e, according to a previous study on diet-related CO2e in Sweden. The participants will be instructed to reduce their consumption of beef and dairy products and increase their consumption of plant-foods i.e. fruits, vegetables, legumes and whole-grain cereals.
  Arms: Climate friendly group
Other: Organic diet — Participants in the 'Organic group' will be assigned an organic diet with very low, or no, content of pesticides. The participants will be instructed to replace at least 50% of their food intake with organic foods.
  Arms: Organic group
Other: Climate friendly and organic diet — The participants in the 'Climate friendly and organic diet group' will be assigned a combination of a climate friendly and organic diet generating low emissions of greenhouse gas and having very low levels of pesticides. The target is to reduce the participants' diet-related CO2e to 2.5 kg per person and day. The participants will be instructed to replace at least 50% of their food intake with organic products.
  Arms: Climate friendly and organic group
Other: Control group (Control diet) — A conventional diet according to the Nordic Nutrition Recommendations (NNR). The participants will get information about the present dietary guidelines and how they can adhere to the guidelines, for example, by implementing the "plate model" for meals and learning about recommended levels of intake of macronutrients, micronutrients, fiber and energy.
  Arms: Control group

SUMMARY:
The aim of this study is to investigate changes in nutrient intake, the human gut microbiota and pesticide excretion in urine when shifting from conventional food habits to sustainable food habits.

ELIGIBILITY:
Inclusion Criteria:

* Living in Västerås
* Carnivores
* Healthy

Exclusion Criteria:

* Vegans

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Changes in composition of the microbiota | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes over time in the presence of all gut bacteria species in the microbiome of the participants based on DNA sequencing from fecal samples. Samples will be collected at three occasions; baseline (reference sample), midtime (after 4 weeks) and at the end (after 8 weeks). From frozen samples, all DNA will be extracted and full shotgun metagenomic sequencing performed using next generation sequencing technologies (Illumina and BGISEQ). A total of 120 samples (3*40 participants) will be sequenced to a depth of at least 3 giga base pairs (Gbp) each.
Changes in concentration of pesticide residues in urine | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in concentration of four pesticide residues (Mepiquat, Chlormequat, Propamocarb and Ethylene thiourea) excreted in urine. Samples will be collected at three occasions; baseline (reference sample), midtime (after 4 weeks) and at the end (after 8 weeks). The concentration of pesticide residues in urine samples will be determined in normal or reversed phase configuration on a high performance liquid chromatograph coupled to a triple quadrupole mass spectrometer (HPLC-MS/MS) system with electrospray ionization interface (ESI) run in negative or positive mode.

SECONDARY OUTCOMES:
Changes in intake of energy | After 8 weeks
  The investigators will assess changes in intake of energy in kilojoule/day (kJ/day) when the participants shifts their diet from conventional food habits to sustainable food habits, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of energy in kJ by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of protein | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of protein in kJ/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of protein in kJ by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of fat | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of fat in kJ/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of fat in kJ by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of carbohydrates | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of carbohydrates in kJ/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of macronutrients in kJ by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of dietary fiber | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of dietary fiber in kJ/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of dietary fiber in kJ by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of vitamin A | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of vitamin A, measured in Retinol Equivalents per day (RE/day), when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin A in RE by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of vitamin D | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of vitamin D, measured in micrograms per day (μg/day), when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin D in μg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of vitamin E | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of vitamin E, measured in alpha-tocopherol equivalents per day (α-TE/day), when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin E in α-TE by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of thiamin | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of thiamin, measured in milligrams per day (mg/day), when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of thiamin in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of riboflavin | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of riboflavin, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of riboflavin in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of niacin | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of niacin, measured in Niacin Equivalents per day (NE/day), when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of niacin in NE by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of vitamin B6 | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of vitamin B6, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin B6 in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of folate | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of folate, measured in μg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of folate in μg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of vitamin B12 | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of vitamin B12, measured in μg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin B12 in μg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of vitamin C | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of vitamin C, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin C in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of calcium | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of calcium, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of calcium in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of phosphorus | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of phosphorus, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of phosphorus in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of potassium | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of potassium, measured in grams per day (g/day), when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of potassium in g by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of iron | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of iron, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of iron in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of zinc | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of zinc, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of zinc in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of iodine | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of iodine, measured in μg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of iodine in μg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of selenium | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of selenium, measured in μg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of selenium in μg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Changes in intake of copper | Baseline, after 4 weeks, after 8 weeks
  The investigators will assess changes in intake of copper, measured in mg/day, when the participants shifts their diet from conventional food habits to sustainable food habits using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of copper in mg by linkage to the National Food Composition Table using the NutriCalc program developed by the research group.
Assessment of the participants likeability of the diets using a questionnaire | After 8 weeks
  The investigators will assess the participants "likeability" of the diets by asking how likely they are to continue to adhere to them after the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Bälter, PhD, Principal Investigator — Mälardalens Högskola
Locations (1):
- Mälardalens University, Västerås, Sweden